CLINICAL TRIAL: NCT01983670
Title: The Investigation of the Pre-movement Facilitation of Agonist-antagonist Muscles and the Effect of the Feedforward Rehabilitation in Individuals With Hypermetria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Associate Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-0951B
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Spinocerebellar Atrophy (SCA)
Keywords: Pre-movement facilitation; Fast goal directed movement; Triphasic EMG pattern; Temporal electrical stimulation,; Spinocerebellar Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- health group 1 (Experimental): Health subjects received 30 mins delay antagonist activation temporal ES.
  Interventions: Other: Temporal electrical stimulation
- SCA group 1 (Experimental): SCA subjects received four weeks temporal ES assisted home training program.
  Interventions: Other: Temporal electrical stimulation
- health group 2 (No Intervention): health subjects controlled group
- SCA group 2 (No Intervention): SCA subjects controlled group

INTERVENTIONS:
Other: Temporal electrical stimulation
  Arms: SCA group 1; health group 1

SUMMARY:
In individuals with spino-cerebellar atrophy (SCA), the delayed onset of antagonist muscle firing has been reported to be the cause of hypermetria. Hypermetria is a common deficit in individuals with spino-cerebellar atrophy SCA when they perform ballistic goal-directed movement. Based on the previous studies, ballistic goal-directed movements are controlled by a triphasic pattern of agonistic and antagonistic muscle activation. The origin of the EMG pattern is a central program, whereas the delayed onset of antagonistic muscle firing has been reported to be the cause of hypermetria. To develop a therapy method, the difference in temporal pattern and intensity of supraspinal excitability of agonist and antagonist bursts between healthy adults and individuals with SCA when performing rapid and slow goal-directed movements should be further investigated.

Traditional rehabilitations of individuals with cerebellum lesion were limited to improve the functional performance of movement. Since the deficits of the goal-directed movement are at pre-movement programming, only feedforward training will be possible to re-establish an appropriate program.

Previous showed that peripheral stimulation resulted in a facilitation of motor cortex. Our group also found that this facilitation in individuals with SCA was similar to the ones without SCA. Therefore, it is possible to adjust the control pattern of supraspinal excitability of agonist and antagonist busts of SCA patient with passively providing electrical stimulation contains normal control pattern of healthy human.

The present study sought to investigate the difference in temporal pattern and intensity of supraspinal excitability of agonist and antagonist bursts between healthy adults and individuals with SCA when performing rapid and slow goal-directed movements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinocerebellar ataxia

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Muscle evoked potential(MEP) | Baseline, 4 weeks.
  Measure of changes in MEP of flexor carpi radialis.
Electromyography(EMG) | Baseline, 4 weeks
  Measure of changes in EMG of flexor carpi radialis and extensor carpi radialis.
Movement error | Baseline, 4weeks
  Measure of changes in movement error during fast 30 degrees wrist extensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Huang YZ, Chang YS, Hsu MJ, Wong AM, Chang YJ. Restoration of Central Programmed Movement Pattern by Temporal Electrical Stimulation-Assisted Training in Patients with Spinal Cerebellar Atrophy. Neural Plast. 2015;2015:462182. doi: 10.1155/2015/462182. Epub 2015 Aug 31. PMID 26417459